CLINICAL TRIAL: NCT05590065
Title: Investigación Clínica Sobre el Impacto en la Seguridad, Viabilidad y Usabilidad de Los Cambios de diseño Realizados en el Dispositivo ABLE Exoskeleton en Pacientes Con lesión Medular en un Entorno Hospitalario
Brief Title: Clinical Investigation on the Impact on Safety, Feasibility and Usability of the Design Changes Performed on ABLE Exoskeleton Device With Spinal Cord Injured Patients in a Hospital Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ABLE Human Motion S.L. (Industry)
Collaborators: Hospital ASEPEYO Sant Cugat (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ABLEexohip; CIV-ES-22-09-040647 (Registry Identifier: EUDAMED)
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Exoskeleton; Robotics; Gait; Rehabilitation; Lower-limb; Neurorehabilitation; Paraplegia; Walking; Assistive technology; Usability; Safety; Feasibility; Multicenter
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 - Treatment (Experimental): Participants with SCI will undergo a training programme with the ABLE Exoskeleton device two times a week for five weeks for a total of 10 sessions.
  Interventions: Device: ABLE Exoskeleton

INTERVENTIONS:
Device: ABLE Exoskeleton — The ABLE Exoskeleton is a lower-limb overground robotic exoskeleton intended for SCI patients for rehabilitation in a clinical setting.

SUMMARY:
The loss of the ability to walk and the associated restriction of mobility presents a major challenge to people with spinal cord injury in an everyday environment designed for pedestrians. Exoskeletal technology has the potential to help people with impaired leg function to regain ambulation and thus improve their independence. This technology is not completely new, but due to their high access price (~120k€/unit), high size and weight (~25 kg), and need for trained physiotherapist supervision, commercially available exoskeletons are only found in large hospitals and only in very few cases get into patients' homes.

The company ABLE Human Motion S.L. (Barcelona, Spain) has developed a novel exoskeleton to overcome these disadvantages, which is more compact, lighter and easier to use.

The primary objective of the study is to investigate the impact of recent design changes performed on the device on the safety, feasibility and usability of the ABLE exoskeleton device in people with spinal cord injury during a five to six weeks gait training programme in a clinical setting. Furthermore, potential effects of the training on walking, general health status, user satisfaction, and quality of life will be assessed.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the impact of the performed design changes on safety, feasibility, and usability of the ABLE Exoskeleton for patients with SCI in a hospital setting during a 5-6 week training programme.

The secondary objectives are as follows:

* Assess the impact of ABLE Exoskeleton training on gait and function.
* Assess the effect on the perceived rate of exertion for patients using the ABLE Exoskeleton.
* Assess the level of user satisfaction from participants and therapists of the ABLE Exoskeleton.

Patients who match inclusion and exclusion criteria and pass pre-study screening will be enrolled in the study. Following the screening, baseline assessments will be conducted without the device. Participants will undergo a training programme with the ABLE Exoskeleton two times a week for five weeks for a total of 10 sessions. Standardized clinical assessments with the device will be performed during the last training sessions. During the training period, several safety and usability measurements will be taken. Two weeks after the final training session a follow-up assessment will be conducted with participants. At the end of the study, the participating therapists will be asked to fill out a satisfaction questionnaire.

The primary hypothesis of this study is that the ABLE Exoskeleton remains safe, feasible, and usable for the intended patient population with SCI in a hospital setting after the implementation of the design changes improving its performance. The secondary hypothesis is that the device will have a positive impact on the perceived rate of exertion, mobility, and level of satisfaction of the study participants with SCI.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age.
* Traumatic and non-traumatic SCI.
* SCI with Neurological Level of Injury (NLI) C5-L5 (from AIS A to AIS D).
* Currently treated as inpatient or outpatient in the investigation center.
* Ability to give informed consent.

Exclusion Criteria:

* WISCI II without exoskeleton of >13
* 5 or more risk factors for fragility as stated by Craven et al (Craven et al., 2009).
* History of lower limb fragility fractures in the last 2 years.
* Deterioration > 3 points of the total International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) motor score within the last 4 weeks.
* Spinal instability.
* Modified Ashworth scale (MAS) of 4 in lower limbs.
* Unable to tolerate 30 min standing without clinical symptoms of orthostatic hypotension
* Psychological or cognitive issues that do not allow a participant to follow the study procedures.
* Known pregnancy or breastfeeding.
* Any neurological condition other than SCI.
* Medically unstable: Unstable CVS, hemodynamic instability, untreated hypertension (SBP>140, DBP>90 mmHg), unresolved DVT, uncontrolled AD.
* Severe comorbidities: any condition that a physician considers to not be appropriate to complete participation in the study.
* Ongoing skin issues: Grade I or higher on EPUAP on areas that will be in contact with exoskeleton (European Pressure Ulcer Advisory Panel, 2019).
* Range of motion (ROM) restrictions in lower extremities, that are incompatible with the device.
* Height, width, weight or other anatomical constraints (such as leg length differences) incompatible with the device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Number and type of Adverse Events [Safety and Tolerability] | Up to 8 weeks
  To assess safety, the number of Severe Adverse Events (SAE), Adverse Events (AE) and drop-outs due to the device will be assessed and reported.
Time and Level of Assistance (LoA) to don/doff the device | Up to 6 weeks
  Level of Assistance (LoA) and time taken to don/doff the device will be measured in every session. LoA will be measured using a 6 item scale, from Total assistance to Independence. Different assistance levels are defined taking into account the degree of participation of both the patient and the therapist on performing the activity.
  This outcome measure will be used to assess the device's usability.
Level of Assistance (LoA) to complete therapy activity tasks | Up to 6 weeks
  Four therapy activity tasks will be attempted every session by the participant. The therapist will record the LoA required to complete each task during the session. The tasks are the following: sit-to-stand, walk 10 meters, turn 180 degrees, and stand-to-sit.
  Different assistance levels are defined taking into account the degree of participation of both the patient and the therapist in performing the activity.
  This outcome measure will be used to assess the device's usability.

SECONDARY OUTCOMES:
BORG Scale | Up to 6 weeks
  Measurement of the perceived rate of exertion. The BORG scale measures the subjective level of intensity in physical work on a 15-grade scale. It will be measured after performing the 6 Minute Walk Test (6 MWT) with the device.
6-Minute Walk Test (6 MWT) | Up to 6 weeks
  6 Minute Walk Test (6 MWT) measures the distance a person can walk in 6 minutes. There are different possibilities for performing this test. For this study, we will use a track of 50 meters, where patients walk back and forth.
10-Meter Walking Test (10 MWT) | Up to 6 weeks
  The 10-Meter Walking Test (10 MWT) measures the time required to walk 10 meters. The test will be performed with a dynamic start with an acceleration distance of 2 meters, a timed 10 meters distance and a deacceleration distance of 2 meters.
Timed up and go test (TUG) | Up to 6 weeks
  Timed Up and Go Test (TUG) measures the time it takes a person to get up from a chair, walk 3 meters, turn around and sit down again. It is a widely used test to assess balance and the risk of falls in different patient groups.
Walking Index for Spinal Cord Injury (WISCI II) | Up to 6 weeks
  WISCI II assesses the extent and nature of assistance for walking 10 meters in persons with SCI. Assistance is specified as different combinations of braces, walking aids and physical assistance. The WISCI II consists of 20 levels from unable to walk to the ability to walk 10 meters without any assistance.
Spinal Cord Independence Measure (SCIM III) | Up to 6 weeks
  SCIM III scale focuses on the ability to perform activities of daily living in persons with SCI. The SCIM III consists of three subscales: Self-Care, Respiratory and Sphincter Management, Mobility (room and toilet) and Mobility (indoors and outdoors, on even surface). A total score of 0 (totally dependent) to 100 (totally independent) points can be achieved.
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) | Up to 6 weeks
  Used to measure user satisfaction from participants and therapists. The Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) is designed to measure the level of satisfaction and the value people attribute to assistive technologies. It does so using 12 variables which are scored on a 5 point scale in terms of perceived importance and satisfaction. While items 1-8 rate the satisfaction with the device, items 9-12 are for assessing the satisfaction with the service. If the users are not very satisfied with a feature, they are asked to provide specific feedback. The final score is the mean sum scores of all valid responses with a range of 1 (not satisfied at all) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Asepeyo Sant Cugat, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porras-Martinez E, Kreamer-Tonin K, Lobo-Prat J, Lopez-Matas H, Carnicero-Carmona A, Tolra-Campanya M, Perez-Canabate F, Estay-Girardi J, Samitier-Pastor B. Enhancing exoskeleton technology through co-creation with clinicians and patients: a pilot study and comparative analysis of the ABLE exoskeleton. Disabil Rehabil. 2025 Nov;47(23):6217-6231. doi: 10.1080/09638288.2025.2496351. Epub 2025 May 7. PMID 40331262